CLINICAL TRIAL: NCT02868229
Title: A Phase 1/2 Randomized, Double-blind, Placebo Controlled, Cohort Dose-escalation Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of COR-001
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of COR-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6018-4791
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COR-001 (Experimental)
  Interventions: Drug: COR-001
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: COR-001
  Arms: COR-001
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial designed to evaluate the safety, pharmacokinetics, and pharmacodynamic effects of multiple doses of COR-001 or placebo

ELIGIBILITY:
INCLUSION CRITERIA

1. Age greater than or equal to 18 years at the time of signing of the ICF.
2. The patient agrees to comply with the contraception and reproduction restrictions of the study
3. Receiving intravenous (IV) or subcutaneous (SC) erythropoietin stimulating agents (ESA) drugs continuously prescribed for a minimum of 8 weeks prior to Screening
4. At least 2 ferritin values during Screening > 300 ng/mL
5. At least 2 transferrin saturation (TSAT) values during Screening between 15% and 50% (inclusive)

EXCLUSION CRITERIA:

1. Use of systemic immunosuppressive drugs during the Screening Period or anticipated use of such drugs any time during the study
2. Clinical evidence or suspicion of active or smoldering infection by clinical or serologic criteria
3. Actively treated or active malignancy
4. Known or suspected occult or active bleeding
5. Received a red blood cell or whole blood transfusion within 2 months prior to Screening or anticipated to receive a blood transfusion at any time during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (12):
- United States (12):
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, North Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Astoria, New York
  - Novo Nordisk Investigational Site, Fresh Meadows, New York
  - Novo Nordisk Investigational Site, Great Neck, New York
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Pergola PE, Devalaraja M, Fishbane S, Chonchol M, Mathur VS, Smith MT, Lo L, Herzog K, Kakkar R, Davidson MH. Ziltivekimab for Treatment of Anemia of Inflammation in Patients on Hemodialysis: Results from a Phase 1/2 Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2021 Jan;32(1):211-222. doi: 10.1681/ASN.2020050595. Epub 2020 Dec 3. PMID 33272965
- [Derived] Pergola PE, Davidson M, Jensen C, Mohseni Zonoozi AA, Raj DS, Andreas Schytz P, Tuttle KR, Perkovic V. Effect of Ziltivekimab on Determinants of Hemoglobin in Patients with CKD Stage 3-5: An Analysis of a Randomized Trial (RESCUE). J Am Soc Nephrol. 2024 Jan 1;35(1):74-84. doi: 10.1681/ASN.0000000000000245. Epub 2023 Dec 13. PMID 38088558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 13 sites in the United States.
Pre-assignment Details: Participants were randomized to ziltivekimab (COR-001) or placebo within each cohort. For the first and other higher dose cohorts, first 2 participants were randomized 1:1 to ziltivekimab or placebo, and were treated at least 48 hours prior to the remaining participants randomized in a 7:1 ratio of ziltivekimab to placebo. For cohorts with doses less than the maximum tolerated dose (MTD) determined from earlier cohorts, randomization was done in 8:2 ratio of ziltivekimab to placebo.
Groups:
- Placebo: Participants received placebo matched to Ziltivekimab once every 14 days for 12 weeks treatment period. Participants were continued on Erythropoiesis stimulating agents (ESA) and parenteral iron, if being given. All the participants were hemodialysis patients.
- COR-001 2 mg: Participants received 2 mg ziltivekimab via Intravenous (IV) infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Randomized participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
- COR-001 6 mg: Participants received 6 mg ziltivekimab via IV infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Randomized participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
- COR-001 20 mg: Participants received 20 mg ziltivekimab via IV infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Randomized participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
Period: Overall Study
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Started | 12 | 16 | 16 | 17
Intent to Treat (ITT) Population | 12 | 16 | 16 | 17
Pharmacodynamic (PD) Population | 12 | 16 | 13 | 12
Pharmacokinetic (PK) Population | 12 | 16 | 16 | 17
Safety Analysis Population | 12 | 16 | 16 | 17
Maximum Tolerated Dose (MTD) Population | 12 | 16 | 16 | 16
Completed | 11 | 16 | 15 | 12
Not Completed | 1 | 0 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Missed dose | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- COR-001 6 mg: Participants received 6 mg ziltivekimab via IV infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
- COR-001 20 mg: Participants received 20 mg ziltivekimab via IV infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
- Total: Total of all reporting groups
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg | Total
Number analyzed (Participants) | 12 | 16 | 16 | 17 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (10.23) | 61.4 (12.95) | 63.8 (10.98) | 57.9 (10.56) | 61.3 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 8 | 9 | 29
  Male | 9 | 7 | 8 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 3 | 4 | 20
  Not Hispanic or Latino | 6 | 9 | 13 | 13 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 10 | 11 | 31
  White | 7 | 10 | 4 | 5 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Characterization of Maximum Tolerated Dose (MTD)
Description: The MTD assessment was based on safety data. If more than 2 of 8 active participants in a cohort experience a Dose-Limiting Toxicities (DLT), the MTD was considered to have been exceeded. The DLT threshold was defined using a threshold of greater than or equal to (>=) Grade 3 events, which includes severe: infusion-related reactions, cardiopulmonary infusion reactions, anaphylaxis, or hypersensitivity.
  DLTs are defined as follows:
  1. Confirmed Grade 3 neutropenia and representing a decline of > 25% from baseline
  2. Serious adverse events (SAEs) of infection in the presence of confirmed Grade 2 or higher new onset lymphopenia or new onset neutropenia.
  3. ≥ Grade 3 ALT (Alanine transaminase) or AST(Aspartate transaminase)
  4. ≥ Grade 4 hematologic toxicity
  5. ≥ Grade 3 non-hematologic toxicity
Time Frame: Weeks 0-24
Population: The MTD analysis population included all participants in the safety analysis population, which included all participants randomized and treated with any amount of study medication with exception of those replaced due to a non-safety reason.
Measure: Number; unit: Events
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Events
  Infection SAEs with confirmed Grade 2 or higher new onset lymphopenia or new onset neutropenia. | 0 | 0 | 0 | 0
  >= Grade 3 ALT or AST | 0 | 0 | 0 | 0
  >= Grade 4 hematologic toxicity | 0 | 0 | 0 | 0
  >= Grade 3 non-hematologic toxicity | 0 | 0 | 0 | 0
  Confirmed Grade 3 neutropenia and representing a decline of > 25% from baseline | 0 | 0 | 0 | 0

2. Primary Outcome: Change in High-sensitivity C-reactive Protein (hsCRP): Week 4
Description: Change from the baseline in hsCRP values to week 4 are presented.
Time Frame: From baseline (mean of screening and day 1) to week 4
Population: The pharmacodynamic (PD) population included all randomized participants who received their assigned study drug, had any PD assessments, and did not have major protocol violations. Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Groups:
- Placebo: Participants received placebo matched to Ziltivekimab once every 14 days for 12 weeks treatment period. Participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients.
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 16 | 11 | 12
Milligrams per liter (mg/L) | 0.373 (3.765) | -10.383 (10.395) | -11.981 (8.232) | -14.561 (11.836)
Statistical Analysis 1: Comparison: Placebo vs COR-001 2 mg; The P-value was obtained from rank transformed analysis of covariance (ANCOVA) model, where the rank transformed change from baseline (CFB) values as the response variable and treatments as a factor and the rank transformed baseline value as its covariate; Test type: Superiority; p = 0.002, ANCOVA; Differences of LS Means = -5.666, 95% CI 2-sided [-9.082 to -2.250]
Statistical Analysis 2: Comparison: Placebo vs COR-001 6 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Differences of LS Means = -6.913, 95% CI 2-sided [-10.613 to -3.214]
Statistical Analysis 3: Comparison: Placebo vs COR-001 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Differences of LS Means = -9.591, 95% CI 2-sided [-13.217 to -5.965]

3. Primary Outcome: Change in Serum Amyloid A (SAA): Week 4
Description: Change from the baseline in serum amyloid A (SAA) values to week 4 are presented.
Time Frame: From baseline (mean of screening and day 1) to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 9 | 16 | 10 | 10
mg/L | -3.733 (6.955) | -22.056 (37.914) | -9.878 (6.687) | -31.910 (41.502)

4. Secondary Outcome: Number of Adverse Events of Special Interest
Description: Frequency of events of interest by treatment group and dose from baseline until the end of the safety follow-up period (week 24) were reported. Adverse events of special interest included severe infusion-related reactions, hypersensitivity reaction during study drug infusion, anaphylaxis and neutropenia events of grade 2 or higher (i.e., absolute neutrophil count <1500/mm^3 and decline by at least 25% from baseline).
Time Frame: Weeks 0-24
Population: The safety analysis population included all participants randomized and treated with any amount of study medication.
Measure: Number; unit: Events
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Events | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An AE (adverse event) is any undesirable event or any untoward medical occurrence that occurs to a participant during the course of a study, or the protocol-defined time after study termination, whether or not that event is considered Study Drug-related. A TEAE was defined as an AE that initiated or worsened on or after the date of first dose of study drug up to the end of study. Number of TEAEs from baseline until the end of safety follow up (week 24) were presented.
Time Frame: Week 0-24
Population: The safety analysis population included all participants randomized and treated with any amount of study medication.
Measure: Number; unit: Events
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Events | 33 | 51 | 83 | 66

6. Secondary Outcome: Electrocardiogram (ECG)
Description: A summary of the overall ECG interpretation and clinical significance from baseline until the end of the safety follow up period (week 24) is presented and categorized as Normal, Abnormal clinically significant (CS), Abnormal non clinically significant (NCS) and Missing.
Time Frame: At baseline, week 6, week 12, week 18 and week 24
Population: The safety analysis population included all participants randomized and treated with any amount of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Participants
  Baseline: Normal | 5 | 7 | 4 | 7
  Baseline: Abnormal, clinically significant (CS) | 1 | 1 | 1 | 1
  Baseline: Abnormal, non clinically significant (NCS) | 6 | 8 | 11 | 9
  Baseline: Missing | 0 | 0 | 0 | 0
  Week 6: Normal | 6 | 3 | 4 | 4
  Week 6: Abnormal, clinically significant (CS) | 1 | 1 | 1 | 0
  Week 6: Abnormal, non clinically significant (NCS) | 5 | 12 | 8 | 10
  Week 6: Missing | 0 | 0 | 3 | 3
  Week 12: Normal | 4 | 5 | 3 | 3
  Week 12: Abnormal, clinically significant (CS) | 1 | 1 | 2 | 1
  Week 12: Abnormal, non clinically significant (NCS) | 7 | 10 | 10 | 11
  Week 12: Missing | 0 | 0 | 1 | 2
  Week 18: Normal | 7 | 4 | 4 | 2
  Week 18: Abnormal, clinically significant (CS) | 1 | 1 | 0 | 0
  Week 18: Abnormal, non clinically significant (NCS) | 4 | 11 | 8 | 9
  Week 18: Missing | 0 | 0 | 4 | 6
  Week 24: Normal | 3 | 5 | 5 | 0
  Week 24: Abnormal, clinically significant (CS) | 1 | 1 | 0 | 1
  Week 24: Abnormal, non clinically significant (NCS) | 7 | 10 | 8 | 10
  Week 24: Missing | 1 | 0 | 3 | 6

7. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies (ADAs)
Description: Number of participants who developed ADAs from baseline until the end of the extended follow up period (week 35) were reported. Samples with detectable ADAs were classified as positive for ADAs. Samples without detectable ADAs were classified as negative for ADAs.
Time Frame: Weeks 0-35
Population: The PK population included all participants who had any valid samples measured for study drug levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Participants
  Positive | 2 | 2 | 1 | 4
  Negative | 10 | 14 | 15 | 13

8. Secondary Outcome: Number of Participants With ADA Titers
Description: Number of participants with ADA titers for ADA-positive samples from baseline to week 35 is presented.
Time Frame: Weeks 0-35
Population: The PK population included all participants who had any valid samples measured for study drug levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Participants | 2 | 2 | 1 | 4

9. Secondary Outcome: Number of Participants With Neutralizing ADAs
Description: Number of participants with neutralizing ADAs from baseline to week 35 are presented.
Time Frame: From baseline (mean of screening and week 1) to week 35
Population: The PK population included all participants who had any valid samples measured for study drug levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 16 | 17
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Transferrin Saturation (TSAT): Week 4
Description: Change from baseline in TSAT to week 4 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of TSAT
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 12 | 12
Percentage of TSAT | 0.467 (6.733) | 5.622 (12.942) | 1.806 (11.197) | 15.778 (12.384)

11. Secondary Outcome: Change in TSAT: Mean of Weeks 10-12
Description: Change from baseline in TSAT to the mean of weeks 10-12 is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of TSAT
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
Percentage of TSAT | 2.278 (8.093) | 6.417 (7.157) | 9.167 (8.569) | 9.028 (6.121)

12. Secondary Outcome: Change in Reticulocyte Hemoglobin (CHr): Week 4
Description: Change from baseline in CHr to week 4 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 16 | 13 | 11
Picograms (pg) | -0.265 (1.216) | 1.197 (1.183) | 1.188 (1.090) | 0.286 (2.265)

13. Secondary Outcome: Change in High Sensitivity C-reactive Protein (Hs-CRP): Mean of 10-12 Weeks
Description: Change from baseline in hs-CRP to the mean of 10-12 weeks is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 12 | 12
mg/L | -0.021 (0.293) | -0.534 (0.439) | -0.916 (0.337) | -1.462 (0.554)

14. Secondary Outcome: Change in SAA: Mean of Weeks 10-12
Description: Change from baseline in SAA to the mean of weeks 10-12 is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
mg/L | -1.262 (19.056) | -24.323 (41.375) | -8.688 (6.665) | -30.324 (37.812)

15. Secondary Outcome: Change in Serum Pre-albumin: Mean of 10-12 Weeks
Description: Change from baseline in serum pre-albumin to the mean of 10-12 weeks is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per decilitre (mg/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
Milligrams per decilitre (mg/dL) | 0.273 (5.716) | 6.032 (6.989) | 8.571 (5.362) | 11.170 (4.983)

16. Secondary Outcome: Change in Albumin: Week 12
Description: Change from baseline in albumin to week 12 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per decilitre (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 11
Grams per decilitre (g/dL) | 0.042 (0.288) | 0.122 (0.212) | 0.192 (0.151) | 0.336 (0.192)

17. Secondary Outcome: Change in Erythropoietin Resistance Index (ERI): Week 4
Description: Change from baseline in ERI to week 4 is presented. ERI is defined as the epoetin alfa-equivalent dose (weight-based per week in U/kg) divided by the serum hemoglobin (in g/dL).
Time Frame: From baseline (weekly mean of screening) to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Unit/kg/week) per (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 16 | 13 | 11
(Unit/kg/week) per (g/dL) | -1.444 (3.590) | -0.975 (1.716) | -3.175 (4.761) | -4.211 (5.785)

18. Secondary Outcome: Change in ERI: Mean of Weeks 8-12
Description: Change from baseline in ERI to the mean of weeks 8-12 is presented. ERI is defined as the epoetin alfa-equivalent dose (weight-based per week in U/kg) divided by the serum hemoglobin (in g/dL).
Time Frame: From baseline (weekly mean of screening), week 8, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Units/kg/week) per (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
(Units/kg/week) per (g/dL) | -2.714 (10.546) | -5.689 (7.824) | -7.842 (8.231) | -8.787 (5.952)

19. Secondary Outcome: Change in ERI: Mean of Weeks 10-12
Description: Change from baseline in ERI to the mean of weeks 10-12 is presented. ERI is defined as the epoetin alfa-equivalent dose (weight-based per week in U/kg) divided by the serum hemoglobin (in g/dL).
Time Frame: From baseline (weekly mean of screening), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Units/kg/week) per (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
(Units/kg/week) per (g/dL) | -2.112 (11.476) | -6.477 (8.756) | -8.272 (8.770) | -8.690 (6.005)

20. Secondary Outcome: Change in CHr: Mean of Weeks 10-12
Description: Change from baseline in CHr to the mean of weeks 10-12 is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
pg | -0.035 (1.264) | 0.859 (1.098) | 1.271 (1.264) | 1.143 (1.635)

21. Secondary Outcome: Change in Hemoglobin: Week 4
Description: Change from baseline in hemoglobin to week 4 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 16 | 13 | 11
g/dL | -0.043 (1.416) | 0.473 (0.751) | 0.805 (0.957) | 0.973 (0.720)

22. Secondary Outcome: Change in Hemoglobin: Mean of Weeks 10-12
Description: Change from baseline in hemoglobin to weeks 10-12 is presented.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
g/dL | -0.107 (1.756) | 0.848 (1.156) | 0.963 (1.131) | 0.772 (1.236)

23. Secondary Outcome: Change in Hemoglobin: Mean of Weeks 10-12, Excluding Hemoglobin Values Following a Change in the Total Weekly ESA Dose
Description: Change from baseline in hemoglobin to weeks 10-12, excluding hemoglobin values following a change in the total weekly ESA (erythropoiesis stimulating agent) dose is presented. A change is defined as the first time when the ESA weekly dose goes up by >25% or down by >25% relative to the previous week's dose.
Time Frame: From baseline (mean of screening and day 1), week 10, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 7 | 6 | 5 | 2
g/dL | 0.352 (1.225) | 0.228 (0.506) | 0.627 (0.988) | 0.567 (1.226)

24. Secondary Outcome: Change in ERI: Week 12
Description: Change from baseline in ERI to week 12 is presented. ERI is defined as the epoetin alfa-equivalent dose (weight-based per week in U/kg) divided by the serum hemoglobin (in g/dL).
Time Frame: From baseline (weekly mean of screening) to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Units/kg/week) per (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 12 | 11
(Units/kg/week) per (g/dL) | -3.229 (12.084) | -6.381 (8.956) | -8.835 (8.785) | -8.690 (6.356)

25. Secondary Outcome: Change in ERI: Mean of Weeks 9-12
Description: Change from baseline in ERI to the mean of weeks 9-12 is presented. ERI is defined as the epoetin alfa-equivalent dose (weight-based per week in U/kg) divided by the serum hemoglobin (in g/dL).
Time Frame: From baseline (weekly mean of screening), week 9, week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Units/kg/week) per (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 12
(Units/kg/week) per (g/dL) | -2.320 (11.392) | -6.338 (8.870) | -8.293 (8.780) | -8.756 (5.949)

26. Secondary Outcome: Change in Hemoglobin: Week 12
Description: Change from baseline in hemoglobin to week 12 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 12 | 11
g/dL | 0.130 (1.240) | 0.502 (1.029) | 0.806 (1.234) | 0.755 (1.379)

27. Secondary Outcome: Change in Hemoglobin: Week 24
Description: Change from baseline in hemoglobin to week 24 is presented.
Time Frame: From baseline (mean of screening and day 1) to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 11 | 8
g/dL | -0.803 (1.929) | 0.154 (1.083) | -0.267 (0.826) | -0.079 (0.703)

28. Secondary Outcome: Change in Hemoglobin From Screening to Peak Hemoglobin: Week 4
Description: Change in hemoglobin from screening to peak hemoglobin at week 4 is presented.
Time Frame: From screening to week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 16 | 13 | 11
g/dL | -0.043 (1.416) | 0.473 (0.751) | 0.805 (0.957) | 0.973 (0.720)

29. Secondary Outcome: Basophils: Week 12
Description: The observed values of basophils at week 12 are presented.
Time Frame: At week 12
Population: The safety analysis population included all participants randomized and treated with any amount of study medication. Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter(10^3 cells/uL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells per microliter(10^3 cells/uL) | 0.03 (0.048) | 0.02 (0.041) | 0.04 (0.051) | 0.03 (0.062)

30. Secondary Outcome: Basophil: Week 24
Description: The observed values of basophils at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
10^3 cells/uL | 0.05 (0.052) | 0.04 (0.062) | 0.08 (0.083) | 0.02 (0.042)

31. Secondary Outcome: Basophils to Leukocytes Ratio: Week 12
Description: Basophils to leukocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of basophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of basophils to leukocytes | 0.65 (0.458) | 0.45 (0.553) | 0.95 (0.447) | 0.87 (0.954)

32. Secondary Outcome: Basophils to Leukocytes Ratio: Week 24
Description: Basophils to leukocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of basophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
Ratio of basophils to leukocytes | 0.62 (0.458) | 0.83 (0.722) | 1.29 (1.296) | 0.57 (0.521)

33. Secondary Outcome: Eosinophils: Week 12
Description: The observed values of eosinophils at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells/uL | 0.16 (0.070) | 0.35 (0.247) | 0.18 (0.080) | 0.65 (1.706)

34. Secondary Outcome: Eosinophils: Week 24
Description: The observed values of eosinophils at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
10^3 cells/uL | 0.19 (0.083) | 0.29 (0.189) | 0.30 (0.336) | 0.36 (0.683)

35. Secondary Outcome: Eosinophils to Leukocytes Ratio: Week 12
Description: Eosinophils to leukocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of eosinophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of eosinophils to leukocytes | 3.39 (1.433) | 5.56 (3.234) | 4.14 (1.669) | 7.32 (10.738)

36. Secondary Outcome: Eosinophils to Leukocytes Ratio: Week 24
Description: The eosinophils to leukocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of eosinophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
Ratio of eosinophils to leukocytes | 3.49 (1.611) | 4.44 (2.287) | 5.32 (4.748) | 3.98 (3.985)

37. Secondary Outcome: Erythrocyte Mean Corpuscular Hemoglobin: Week 12
Description: The observed values of erythrocyte mean corpuscular hemoglobin at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
pg | 30.2 (1.48) | 31.3 (2.66) | 30.8 (2.15) | 31.2 (2.48)

38. Secondary Outcome: Erythrocyte Mean Corpuscular Hemoglobin: Week 24
Description: The observed values of erythrocyte mean corpuscular hemoglobin at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
pg | 29.5 (2.54) | 31.0 (2.80) | 30.6 (2.40) | 29.6 (2.46)

39. Secondary Outcome: Erythrocyte Mean Corpuscular Hemoglobin (HGB) Concentration: Week 12
Description: The observed values of erythrocyte mean corpuscular HGB concentration at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Grams per deciliter (g/dL) | 30.86 (1.332) | 31.41 (1.438) | 29.75 (1.563) | 31.23 (0.978)

40. Secondary Outcome: Erythrocyte Mean Corpuscular HGB Concentration: Week 24
Description: The observed values of erythrocyte mean corpuscular HGB concentration at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
g/dL | 30.78 (1.572) | 31.04 (1.307) | 29.52 (1.799) | 30.28 (1.297)

41. Secondary Outcome: Erythrocyte Mean Corpuscular Volume: Week 12
Description: The observed values of erythrocyte mean corpuscular volume at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
femtoliters (fL) | 98.16 (4.328) | 99.35 (6.923) | 103.49 (9.153) | 99.97 (8.089)

42. Secondary Outcome: Erythrocyte Mean Corpuscular Volume: Week 24
Description: The observed values of erythrocyte mean corpuscular volume at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
fL | 95.70 (6.096) | 99.69 (6.859) | 103.53 (8.550) | 97.76 (6.983)

43. Secondary Outcome: Erythrocytes: Week 12
Description: The observed values of erythrocytes at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter(10^6 cells/uL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^6 cells per microliter(10^6 cells/uL) | 3.464 (0.302) | 3.348 (0.438) | 3.459 (0.411) | 3.370 (0.345)

44. Secondary Outcome: Erythrocytes: Week 24
Description: The observed values of erythrocytes at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^6 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
10^6 cells/uL | 3.312 (0.480) | 3.256 (0.347) | 3.111 (0.388) | 3.365 (0.513)

45. Secondary Outcome: Hematocrit: Week 12
Description: The observed values of hematocrit at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage of Hematocrit
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Percentage of Hematocrit | 34.0 (3.43) | 33.1 (3.31) | 35.6 (3.13) | 33.7 (4.24)

46. Secondary Outcome: Hematocrit: Week 24
Description: The observed values of hematocrit at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage of Hematocrit
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
Percentage of Hematocrit | 31.5 (3.72) | 32.4 (2.78) | 32.2 (4.11) | 32.8 (3.58)

47. Secondary Outcome: Hemoglobin: Week 12
Description: The observed values of hemoglobin at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
g/dL | 10.51 (1.190) | 10.37 (0.928) | 10.56 (1.018) | 10.53 (1.360)

48. Secondary Outcome: Hemoglobin: Week 24
Description: The observed values of hemoglobin at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
g/dL | 9.68 (1.057) | 10.06 (1.031) | 9.47 (1.135) | 9.87 (1.215)

49. Secondary Outcome: Hypochromatic Red Cells Week 12
Description: The observed values of hypochromatic red cells at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage of Hypochromatic red cells
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Percentage of Hypochromatic red cells | 13.65 (15.015) | 12.09 (11.191) | 23.65 (22.214) | 11.99 (14.657)

50. Secondary Outcome: Hypochromatic Red Cells: Week 24
Description: The observed values of hypochromatic red cells at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage of Hypochromatic red cells
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
Percentage of Hypochromatic red cells | 11.88 (10.819) | 11.60 (11.895) | 32.02 (25.224) | 15.44 (13.415)

51. Secondary Outcome: Leukocytes: Week 12
Description: The observed values of leukocytes at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells/uL | 5.23 (1.718) | 5.84 (1.837) | 4.68 (1.069) | 5.25 (3.004)

52. Secondary Outcome: Leukocytes: Week 24
Description: The observed values of leukocytes at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
10^3 cells/uL | 5.52 (2.197) | 6.06 (1.689) | 5.52 (1.168) | 6.13 (3.414)

53. Secondary Outcome: Lymphocytes: Week 12
Description: The observed values of lymphocytes at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells/uL | 1.10 (0.306) | 1.45 (0.678) | 1.11 (0.250) | 1.18 (0.388)

54. Secondary Outcome: Lymphocytes: Week 24
Description: The observed values of lymphocytes at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
10^3 cells/uL | 1.10 (0.452) | 1.26 (0.496) | 1.08 (0.267) | 1.23 (0.523)

55. Secondary Outcome: Lymphocytes to Leukocytes Ratio: Week 12
Description: Lymphocytes to leukocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of lymphocytes to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of lymphocytes to leukocytes | 22.86 (9.139) | 25.09 (9.611) | 24.15 (5.774) | 24.81 (7.341)

56. Secondary Outcome: Lymphocytes to Leukocytes Ratio at Week 24
Description: Lymphocytes to leukocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of lymphocytes to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
Ratio of lymphocytes to leukocytes | 21.47 (11.350) | 21.24 (7.195) | 20.63 (6.997) | 21.71 (7.633)

57. Secondary Outcome: Monocytes: Week 12
Description: The observed values of monocytes at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells/uL | 0.26 (0.151) | 0.29 (0.171) | 0.25 (0.102) | 0.31 (0.119)

58. Secondary Outcome: Monocytes: Week 24
Description: The observed values of monocytes at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
10^3 cells/uL | 0.40 (0.184) | 0.39 (0.200) | 0.31 (0.138) | 0.30 (0.067)

59. Secondary Outcome: Monocytes to Leukocytes Ratio: Week 12
Description: Monocytes to leukocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of monocytes to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of monocytes to leukocytes | 5.61 (2.871) | 5.42 (2.649) | 5.15 (1.652) | 6.21 (2.230)

60. Secondary Outcome: Monocytes to Leukocytes Ratio: Week 24
Description: Monocytes to leukocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of monocytes to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
Ratio of monocytes to leukocytes | 7.04 (2.369) | 6.29 (2.281) | 5.49 (1.770) | 5.77 (2.396)

61. Secondary Outcome: Neutrophils: Week 12
Description: The observed values of neutrophils at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
10^3 cells/uL | 3.68 (1.611) | 3.70 (1.455) | 3.09 (0.921) | 3.09 (1.354)

62. Secondary Outcome: Neutrophils: Week 24
Description: The observed values of neutrophils at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
10^3 cells/uL | 3.82 (1.795) | 4.08 (1.252) | 3.71 (1.047) | 4.25 (2.507)

63. Secondary Outcome: Neutrophils to Leukocytes Ratio: Week 12
Description: Neutrophils to leukocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of neutrophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of neutrophils to leukocytes | 67.29 (11.707) | 62.41 (10.148) | 65.61 (7.447) | 60.79 (9.656)

64. Secondary Outcome: Neutrophils to Leukocytes Ratio: Week 24
Description: Neutrophils to leukocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of neutrophils to leukocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 10
Ratio of neutrophils to leukocytes | 67.37 (13.396) | 67.21 (8.771) | 67.31 (8.293) | 67.94 (8.750)

65. Secondary Outcome: Platelets: Week 12
Description: The observed values of platelets at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 14
10^3 cells/uL | 169.8 (68.37) | 168.3 (38.62) | 129.4 (42.26) | 143.8 (48.68)

66. Secondary Outcome: Platelets: Week 24
Description: The observed values of platelets at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
10^3 cells/uL | 180.2 (62.44) | 203.1 (57.78) | 151.6 (41.75) | 160.1 (55.67)

67. Secondary Outcome: Reticulocytes to Erythrocytes Ratio: Week 12
Description: Reticulocytes to erythrocytes ratio at week 12 is presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of reticulocytes to erythrocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 10 | 15 | 14 | 15
Ratio of reticulocytes to erythrocytes | 1.92 (0.852) | 1.68 (0.757) | 2.14 (1.203) | 2.32 (1.537)

68. Secondary Outcome: Reticulocytes to Erythrocytes Ratio: Week 24
Description: Reticulocytes to erythrocytes ratio at week 24 is presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Ratio of reticulocytes to erythrocytes
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 10
Ratio of reticulocytes to erythrocytes | 1.95 (0.872) | 1.96 (0.669) | 1.84 (0.612) | 2.24 (0.935)

69. Secondary Outcome: Alanine Aminotransferase: Week 12
Description: The observed values of alanine aminotransferase at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
units per liter (U/L) | 12.1 (6.61) | 18.6 (13.85) | 19.9 (10.89) | 19.0 (9.43)

70. Secondary Outcome: Alanine Aminotransferase: Week 24
Description: The observed values of alanine aminotransferase at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
U/L | 8.7 (4.67) | 11.9 (4.78) | 15.3 (6.81) | 15.4 (6.35)

71. Secondary Outcome: Albumin: Week 12
Description: The observed values of albumin at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
g/dL | 3.96 (0.382) | 3.90 (0.210) | 3.97 (0.304) | 3.98 (0.273)

72. Secondary Outcome: Albumin: Week 24
Description: The observed values of albumin at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
g/dL | 3.75 (0.432) | 3.83 (0.305) | 3.77 (0.347) | 3.84 (0.456)

73. Secondary Outcome: Alkaline Phosphatase: Week 12
Description: The observed values of alkaline phosphatase at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
U/L | 103.0 (56.43) | 125.4 (87.32) | 107.5 (57.54) | 106.2 (44.69)

74. Secondary Outcome: Alkaline Phosphatase: Week 24
Description: The observed values of alkaline phosphatase at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
U/L | 99.8 (51.17) | 140.6 (119.26) | 121.2 (55.26) | 95.2 (53.01)

75. Secondary Outcome: Aspartate Aminotransferase: Week 12
Description: The observed values of aspartate aminotransferase at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
U/L | 15.5 (5.89) | 18.1 (11.57) | 20.5 (10.85) | 15.7 (4.61)

76. Secondary Outcome: Aspartate Aminotransferase: Week 24
Description: The observed values of aspartate aminotransferase at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
U/L | 14.7 (5.57) | 14.3 (5.59) | 17.3 (7.75) | 14.7 (3.20)

77. Secondary Outcome: Bicarbonate: Week 12
Description: The observed values of bicarbonate at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
millimoles per liter (mmol/L) | 23.5 (3.06) | 23.1 (3.03) | 22.7 (3.26) | 25.5 (3.50)

78. Secondary Outcome: Bicarbonate: Week 24
Description: The observed values of bicarbonate at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mmol/L | 23.3 (3.00) | 24.6 (2.83) | 22.4 (2.43) | 26.0 (3.28)

79. Secondary Outcome: Bilirubin: Week 12
Description: The observed values of bilirubin at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 0.490 (0.186) | 0.450 (0.157) | 0.603 (0.234) | 0.553 (0.150)

80. Secondary Outcome: Bilirubin: Week 24
Description: The observed values of bilirubin at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 0.450 (0.169) | 0.430 (0.142) | 0.565 (0.184) | 0.520 (0.125)

81. Secondary Outcome: Calcium: Week 12
Description: The observed values of calcium at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 8.89 (0.883) | 8.54 (0.737) | 8.90 (0.777) | 8.39 (0.727)

82. Secondary Outcome: Calcium: Week 24
Description: The observed values of calcium at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 8.73 (0.740) | 8.95 (0.734) | 8.76 (0.653) | 8.82 (1.011)

83. Secondary Outcome: Chloride: Week 12
Description: The observed values of chloride at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mmol/L | 97.0 (3.69) | 98.6 (5.34) | 98.0 (4.87) | 98.5 (2.47)

84. Secondary Outcome: Chloride: Week 24
Description: The observed values of chloride at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mmol/L | 98.5 (3.67) | 97.7 (4.76) | 98.7 (3.15) | 97.6 (3.73)

85. Secondary Outcome: Cholesterol: Week 12
Description: The observed values of cholesterol at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 140.4 (41.24) | 140.3 (40.51) | 145.9 (41.38) | 146.0 (43.54)

86. Secondary Outcome: Cholesterol: Week 24
Description: The observed values of cholesterol at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 130.5 (40.19) | 148.3 (38.74) | 131.2 (36.17) | 158.0 (44.04)

87. Secondary Outcome: Creatinine: Week 12
Description: The observed values of creatinine at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 9.458 (2.739) | 9.616 (2.642) | 9.227 (2.526) | 10.115 (3.391)

88. Secondary Outcome: Creatinine: Week 24
Description: The observed values of creatinine at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 9.086 (2.260) | 9.173 (2.541) | 9.027 (2.216) | 9.703 (3.714)

89. Secondary Outcome: Direct Bilirubin: Week 12
Description: The observed values of direct bilirubin at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 0.101 (0.071) | 0.098 (0.066) | 0.123 (0.049) | 0.118 (0.059)

90. Secondary Outcome: Direct Bilirubin: Week 24
Description: The observed values of direct bilirubin at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 0.105 (0.081) | 0.081 (0.046) | 0.124 (0.053) | 0.102 (0.042)

91. Secondary Outcome: Glucose: Week 12
Description: The observed values of glucose at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 123.1 (52.29) | 128.5 (66.17) | 119.6 (73.49) | 101.2 (19.86)

92. Secondary Outcome: Glucose: Week 24
Description: The observed values of glucose at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 129.5 (54.83) | 129.9 (64.12) | 142.4 (168.55) | 104.2 (22.97)

93. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol: Week 12
Description: The observed values of HDL cholesterol at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 51.6 (16.47) | 50.1 (18.05) | 54.2 (17.17) | 52.5 (15.14)

94. Secondary Outcome: HDL Cholesterol: Week 24
Description: The observed values of HDL cholesterol at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 50.5 (17.33) | 45.4 (16.02) | 48.8 (16.29) | 46.8 (22.49)

95. Secondary Outcome: Hepcidin-25: Week 12
Description: The observed values of hepcidin-25 at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 13 | 14
nanogram/milliliter (ng/mL) | 310.67 (163.569) | 344.99 (154.189) | 288.72 (210.049) | 233.89 (114.748)

96. Secondary Outcome: Hepcidin-25: Week 24
Description: The observed values of hepcidin-25 at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
ng/mL | 347.55 (167.752) | 328.35 (159.543) | 302.72 (131.966) | 262.18 (118.461)

97. Secondary Outcome: Low-density Lipoproteins (LDL) Cholesterol: Week 12
Description: The observed values of LDL cholesterol at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 15 | 15 | 15
mg/dL | 67.2 (29.62) | 61.4 (31.40) | 63.8 (32.69) | 68.1 (39.58)

98. Secondary Outcome: LDL Cholesterol: Week 24
Description: The observed values of LDL cholesterol at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 12
mg/dL | 60.9 (32.59) | 69.4 (30.44) | 54.7 (27.73) | 82.7 (35.43)

99. Secondary Outcome: Lipoprotein-a: Week 12
Description: The observed values of lipoprotein-a at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Nanomoles per litre (nmol/L)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
Nanomoles per litre (nmol/L) | 35.2 (38.88) | 86.3 (83.29) | 68.9 (50.11) | 53.1 (41.54)

100. Secondary Outcome: Lipoprotein-a: Week 24
Description: The observed values of lipoprotein-a at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
nmol/L | 39.3 (37.60) | 96.6 (92.52) | 89.5 (61.25) | 61.9 (52.28)

101. Secondary Outcome: Phosphate: Week 12
Description: The observed values of phosphate at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 5.06 (1.425) | 5.67 (1.905) | 6.51 (1.364) | 5.43 (1.416)

102. Secondary Outcome: Phosphate: Week 24
Description: The observed values of phosphate at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 5.55 (1.841) | 4.57 (1.399) | 5.15 (0.724) | 5.64 (1.459)

103. Secondary Outcome: Potassium: Week 12
Description: The observed values of potassium at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mmol/L | 5.13 (1.094) | 5.06 (0.754) | 5.03 (0.662) | 4.69 (0.647)

104. Secondary Outcome: Potassium: Week 24
Description: The observed values of potassium at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mmol/L | 4.96 (0.628) | 4.97 (0.581) | 4.71 (0.466) | 4.75 (0.762)

105. Secondary Outcome: Sodium: Week 12
Description: The observed values of sodium at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mmol/L | 135.8 (2.80) | 137.1 (4.55) | 137.4 (4.03) | 138.6 (3.64)

106. Secondary Outcome: Sodium: Week 24
Description: The observed values of sodium at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mmol/L | 136.7 (3.04) | 136.2 (4.90) | 137.8 (4.24) | 137.2 (4.06)

107. Secondary Outcome: Triglycerides: Week 12
Description: The observed values of triglyceride at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 107.9 (50.59) | 140.8 (131.19) | 139.5 (85.00) | 126.7 (89.04)

108. Secondary Outcome: Triglycerides: Week 24
Description: The observed values of triglycerides at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 95.4 (53.98) | 166.9 (120.39) | 146.6 (147.52) | 142.9 (95.94)

109. Secondary Outcome: Urea Nitrogen: Week 12
Description: The observed values of urea nitrogen at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 15
mg/dL | 61.7 (26.03) | 61.1 (17.40) | 53.3 (12.38) | 62.1 (21.06)

110. Secondary Outcome: Urea Nitrogen: Week 24
Description: The observed values of urea nitrogen at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mg/dL | 66.2 (30.04) | 59.9 (16.97) | 51.1 (13.67) | 59.6 (15.11)

111. Secondary Outcome: Pre-dialysis Body Mass Index (BMI): Week 12
Description: Pre-dialysis BMI values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: kilogram per meter^2 (kg/m^2)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
kilogram per meter^2 (kg/m^2) | 28.952 (5.774) | 29.668 (8.674) | 32.150 (9.365) | 32.574 (8.240)

112. Secondary Outcome: Pre-infusion BMI: Week 11
Description: Pre-infusion BMI values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 9 | 9 | 7 | 6
Kg/m^2 | 29.337 (6.800) | 29.399 (8.267) | 31.290 (8.341) | 34.163 (7.950)

113. Secondary Outcome: Pre-dialysis Diastolic Blood Pressure: Week 12
Description: Pre-dialysis diastolic blood pressure values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mm Hg)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
Millimetre of mercury (mm Hg) | 84.8 (21.14) | 70.4 (11.70) | 84.2 (10.23) | 76.3 (16.29)

114. Secondary Outcome: Pre-dialysis Diastolic Blood Pressure: Week 24
Description: Pre-dialysis diastolic blood pressure values at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mm Hg | 76.9 (13.59) | 77.8 (13.23) | 74.0 (14.53) | 78.8 (13.74)

115. Secondary Outcome: Pre-infusion Diastolic Blood Pressure: Week 11
Description: Pre-infusion diastolic blood pressure values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 15 | 12
mm Hg | 82.3 (19.68) | 66.6 (10.03) | 75.8 (11.80) | 78.7 (10.71)

116. Secondary Outcome: Pre-dialysis Heart Rate: Week 12
Description: Pre-dialysis heart rate values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
beats/min | 69.3 (7.50) | 71.1 (12.20) | 70.8 (8.03) | 76.9 (13.37)

117. Secondary Outcome: Pre-dialysis Heart Rate: Week 24
Description: Pre-dialysis heart rate values at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
beats/min | 71.8 (12.02) | 78.0 (11.90) | 72.6 (10.03) | 78.9 (17.72)

118. Secondary Outcome: Pre-infusion Heart Rate: Week 11
Description: Pre-infusion heart rate values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 15 | 12
beats/min | 67.1 (6.11) | 70.1 (9.44) | 65.7 (8.88) | 72.8 (9.80)

119. Secondary Outcome: Pre-dialysis Respiration Rate: Week 12
Description: Pre-dialysis respiration rate values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
breaths per minute (breaths/min) | 17.8 (1.27) | 17.9 (1.29) | 17.9 (1.53) | 18.1 (1.31)

120. Secondary Outcome: Pre-dialysis Respiration Rate: Week 24
Description: Pre-dialysis respiration rate values at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 12 | 12
breaths/min | 16.6 (2.69) | 18.1 (1.09) | 18.3 (1.60) | 18.4 (1.08)

121. Secondary Outcome: Pre-infusion Respiration Rate: Week 11
Description: Pre-infusion respiration rate values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 15 | 12
breaths/min | 18.1 (1.22) | 17.8 (1.24) | 18.1 (1.39) | 18.3 (1.23)

122. Secondary Outcome: Pre-dialysis Systolic Blood Pressure: Week 12
Description: Pre-dialysis values of systolic blood pressure at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
mm Hg | 164.4 (33.13) | 143.8 (21.04) | 164.3 (25.17) | 151.4 (26.83)

123. Secondary Outcome: Pre-dialysis Systolic Blood Pressure: Week 24
Description: Pre-dialysis values of systolic blood pressure at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
mm Hg | 149.4 (30.43) | 146.7 (19.14) | 157.6 (27.45) | 155.8 (22.93)

124. Secondary Outcome: Pre-infusion Systolic Blood Pressure: Week 11
Description: Pre-infusion systolic blood pressure values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 15 | 12
mm Hg | 161.2 (25.78) | 138.7 (27.32) | 144.0 (28.30) | 152.1 (28.18)

125. Secondary Outcome: Pre-dialysis Weight: Week 12
Description: Pre-dialysis weight values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
Kilogram (Kg) | 84.583 (18.464) | 82.162 (28.830) | 92.120 (25.720) | 96.213 (29.206)

126. Secondary Outcome: Pre-infusion Weight: Week 11
Description: Pre-infusion weight values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 9 | 9 | 7 | 6
Kg | 86.356 (21.881) | 83.433 (31.580) | 92.043 (26.401) | 91.217 (15.121)

127. Secondary Outcome: Pre-dialysis Temperature: Week 12
Description: Pre-dialysis temperature values at week 12 are presented.
Time Frame: At week 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 12 | 16 | 15 | 16
Celsius (C) | 36.259 (0.572) | 36.435 (0.304) | 36.436 (0.314) | 36.490 (0.157)

128. Secondary Outcome: Pre-dialysis Temperature: Week 24
Description: Pre-dialysis temperature values at week 24 are presented.
Time Frame: At week 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 13 | 12
C | 36.328 (0.384) | 36.440 (0.315) | 36.168 (0.370) | 36.361 (0.251)

129. Secondary Outcome: Pre-infusion Temperature: Week 11
Description: Pre-infusion temperature values at week 11 are presented.
Time Frame: At week 11
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 11 | 16 | 15 | 12
C | 36.182 (0.692) | 36.377 (0.259) | 36.187 (0.494) | 36.375 (0.193)

130. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time 0 to Infinity (AUC 0-α) of COR-001
Description: Area under the serum concentration time curve from time 0 to infinity (AUC 0-α) of COR-001 is presented.
Time Frame: Week 1 (day 1, 3, and 5), Week 2 (day 8), Week 3 (day 15), Week 5 (day 29), Week 7 (day 43), Week 8 (day 50), Week 9 (day 57), Week 11 (day 71 and 75), Week 14 (day 92), Week 18 (day 120) and Week 35 (day 239).
Population: The PK population included all participants who had any valid samples measured for study drug levels. Overall number of participants analysed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: nanogram*day/milliliter (ng*day/mL)
Arm/Group | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 16 | 14 | 14
nanogram*day/milliliter (ng*day/mL) | 11962 (4731) | 40911 (23629) | 118177 (60393)

131. Secondary Outcome: Elimination Half-life in the Initial Phase (t 1/2,α)
Description: Elimination half-life in the initial phase (t 1/2,α) is presented from week 0 to week 35.
Time Frame: as for outcome 130
Population: as for outcome 130
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 16 | 14 | 14
Days | 2.55 (0.94) | 1.98 (0.87) | 1.90 (0.70)

132. Secondary Outcome: Elimination Half-life in the Terminal Phase (t 1/2, z)
Description: Elimination half-life in the terminal phase(t 1/2, z) is presented from week 0 to week 35.
Time Frame: as for outcome 130
Population: as for outcome 130
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 16 | 14 | 14
Days | 51.44 (21.55) | 38.22 (14.21) | 40.93 (13.43)

133. Secondary Outcome: Maximum Serum Concentration (Cmax)
Description: Maximum serum concentration (Cmax) of COR-001 from week 0 to week 35 is presented.
Time Frame: as for outcome 130
Population: as for outcome 130
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
Number analyzed (Participants) | 16 | 14 | 14
ng/mL | 378 (93) | 1368 (359) | 3584 (1349)

134. Secondary Outcome: Impact of ADAs on Pharmacokinetics
Description: Presence of ADA was a covariate for pharmacokinetics (PK) affecting V1 (volume of distribution for the central compartment). Impact of ADAs on V1 from baseline to week 35 is presented. In the below table, result presented is the bootstrap parameter estimate of the effect of ADA on V1 for a PK model that includes data for all arms combined.
Time Frame: as for outcome 130
Population: as for outcome 130
Measure: Mean (95% Confidence Interval); unit: Milliliter (mL)
Groups:
- COR-001: Participants were randomized to ziltivekimab (COR-001) or placebo within each cohort. Participants received 2 mg or 6 mg or 20 mg ziltivekimab via IV infusion once every 14 days over approximately 60 minutes, which started any time prior to the last 1 hour of dialysis for 12 weeks treatment period. Randomized participants were continued on ESA and parenteral iron, if being given. All the participants were hemodialysis patients
Arm/Group | COR-001
Number analyzed (Participants) | 61
Milliliter (mL) | 0.361 [0.0548 to 0.658]

ADVERSE EVENTS:
Time Frame: Weeks 0-24
Description: All presented AEs are TEAEs. A treatment-emergent adverse event (TEAE) was defined as an AE that initiated or worsened on or after the date of first dose of study drug up to the end of the study.The results are based on the safety analysis set which included all patients randomized and treated with any amount of study medication.
Arm/Group | Placebo | COR-001 2 mg | COR-001 6 mg | COR-001 20 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16 | 2/16 | 2/17
Serious Adverse Events (participants affected / at risk) | 3/12 | 4/16 | 7/16 | 6/17
Other Adverse Events (participants affected / at risk) | 7/12 | 11/16 | 15/16 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | COR-001 2 mg (N=16) | COR-001 6 mg (N=16) | COR-001 20 mg (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dialysis disequilibrium syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | COR-001 2 mg (N=16) | COR-001 6 mg (N=16) | COR-001 20 mg (N=17)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial conduction time prolongation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 4 (5) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iris neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02868229/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT02868229/SAP_001.pdf